CLINICAL TRIAL: NCT03321994
Title: A Single-center, Randomized, Active-controlled and Evaluator-blind Investigator-initiated Trial to Evaluate and Compare the Efficacy and Safety of CT-guided Needle Guidance Using Stereotaxic Unit, Navigation Versus Conventional Biopsy Technique for the Patients Scheduled to Undergo Percutaneous Pulmonary Nodule Biopsy
Brief Title: CT-guided Needle Guidance Using Stereotaxic Unit, Navigation Versus Conventional Biopsy Technique for the Percutaneous Pulmonary Nodule Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hyung Jin Won (Other)
Responsible Party: Sponsor-Investigator, Hyung Jin Won, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AS-NPR-03
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Percutaneous Pulmonary Nodule Biopsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotaxic unit, navigation (Experimental)
  Interventions: Device: stereotaxic unit, navigation
- Conventional biopsy technique (Active Comparator)
  Interventions: Device: conventional biopsy technique

INTERVENTIONS:
Device: stereotaxic unit, navigation — CT-guided needle guidance using stereotaxic unit, navigation
  Arms: Stereotaxic unit, navigation
Device: conventional biopsy technique — CT-guided needle guidance using conventional biopsy technique
  Arms: Conventional biopsy technique

SUMMARY:
The purpose of this study was to compare the safety and efficacy of CT-guided needle guidance using stereotaxic unit, navigation versus conventional biopsy technique for the patients scheduled to undergo percutaneous pulmonary nodule biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with localized lesions such as pulmonary nodules on chest x-ray, CT or PET CT
* Histopathologic examination is necessary if lung lesion is unknown
* Histologic findings affect the disease stage or treatment plan
* If the investigator decides to perform a percutaneous lung biopsy because the biopsy or diagnosis through the bronchoscopy is not possible or has low risk-benefit
* Patient who have consented to contraception during the period of clinical trial participation (one month after the procedure)
* Patient who voluntarily agree to participate in this clinical trial and are willing to comply with the protocol

Exclusion Criteria:

* Patient with pulmonary function insufficiency
* Patient who has difficulty in self-breathing (e.g, breathing through oxygen breathing apparatus)
* Patient with Uncontrolled coagulation disorders (INR > 1.3 or Blood platelet count < 50,000/µl)
* Patient with allergy to CT contrast agent
* Patient under 19 years old or over 80 years old
* Pregnant or lactating
* Patient with uncontrollable systemic disease (e.g, uncontrolled hypertension, uncontrolled cardiovascular disease, etc.)
* Patient who currently participating or has participated in other clinical trials within 30 days of the screening date
* If it is judged inappropriate to participate in this clinical trial under the judgment of the investigator

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Needle guide accuracy(mm) | 1 day
  3D distance between target point and actual needle tip

SECONDARY OUTCOMES:
Needle guide angle deviation(°) | 1 day
  The angle deviation between the needle insertion path on the procedure plan and the path of the actually inserted needle
Number of needle readjustments | 1 day
  Retract the inserted needle and adjust the direction
Number of needle reinsertion | 1 day
  Needle is completely pulled out and then inserted again
Needle insertion time(min) | 1 day
  Time from pre-CT scan to the last CT scan before lung biopsy
Procedure time(min) | 1 day
  Time from pre-CT scan to dressing after lung biopsy

OTHER OUTCOMES:
Radiation dose(DLP, mGy·cm) | 1 day
  DLP(mGy·cm) = CTDIvol x scan length
Occurrence rate of adverse device effect(%) | 1 month
  Adverse events that are correlated with the needle insertion procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Jin Won, MD., PhD, Principal Investigator — Asan Medical Center, Seoul, Korea